CLINICAL TRIAL: NCT03617562
Title: Arthroscopic Partial Repair vs. Superior Capsular Reconstruction for Massive Irreparable Rotator Cuff Tears: A Pilot Randomized and Controlled Trial
Brief Title: Superior Capsular Reconstruction vs. Partial Repair for Massive Rotator Cuff Tears
Acronym: SCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Women's College Hospital (Other); St. Joseph's Healthcare Hamilton (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCR2018
Record Dates: First submitted 2018-05-07; First posted 2018-08-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Rotator Cuff Tear
Keywords: Massive Rotator Cuff Tear; Shoulder Injuries
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Superior Capsular Reconstruction (Experimental): Patients will be treated with the new technique of superior capsular reconstruction with dermal allograft.
  Interventions: Procedure: Superior Capsular Reconstruction
- Partial Repair (Active Comparator): Patients will have a partial repair with residual defect as an established standard procedure.
  Interventions: Procedure: Partial Repair

INTERVENTIONS:
Procedure: Superior Capsular Reconstruction — Residual rotator cuff defect is reconstructed with a dermal allograft secured to the glenoid and humeral head.
  Arms: Superior Capsular Reconstruction
Procedure: Partial Repair — Rotator cuff is repaired with residual defect remaining.
  Arms: Partial Repair

SUMMARY:
Little evidence exists to guide treatment in patients with massive irreparable rotator cuff tears (MRCTS). Arthroscopic partial rotator cuff repair (PRCR) has the longest record of use. The new technique of superior capsular reconstruction (SCR) has more recently been described. Despite high enthusiasm for this technique, its effectiveness, cost and safety profile have not been established.

The long-term goal of this study is to perform a multicenter randomized control trial to evaluate the effectiveness of SCR compared to PRCR in patients with MRCTS. The current study is a pilot required to support the development of an expanded formal clinical trial.

DETAILED DESCRIPTION:
The current study seeks to improve the management of patients suffering from massive irreparable rotator cuff tears. Despite several available surgical options, no level 1 evidence or randomized clinical trials have been performed in this patient population to date. Arthroscopic partial rotator cuff repair (PRCR) is arguably the gold-standard surgical option with the longest record of use. The new technique of superior capsular reconstruction (SCR) has also emerged with early biomechanical and case series showing promising results. SCR has quickly made its way into clinical practice in North America. Despite this, the effectiveness, cost, and safety profile has not been established for this procedure. As such, patients with massive irreparable rotator cuff tears are in need of high level evidence to support surgical decision making, particular with regards to the proliferation of SCR surgery.

This pilot study is a randomized, controlled, double-blinded trial comparing superior capsular reconstruction using dermal allograft with arthroscopic partial repair in patients with massive irreparable rotator cuff tears. In this study, "double-blind" includes study patients and outcome assessors. Randomization will occur intra-operatively once a tear is determined to be irreparable.

This trial will be conducted at 7 sites and involve 7 surgeons. Surgeons must meet eligibility requirements to participate (shoulder or sports fellowship-trained, minimum of 3 SCR procedures, and 25 arthroscopic rotator cuff repair procedures in the past year). A member of the local research team will pre-screen consults of eligible patients. Full eligibility will be determined during the primary appointment with an orthopaedic surgeon. Baseline data will be recorded following informed consent. Postoperative outcomes will be measured during regularly scheduled clinic visits (6 weeks, 3 months, 6 months, 1-year and 2-year post-surgery).

Prior to surgery, patients will have informed consent for both procedures, with randomization to be performed intraoperatively. Based on initial arthroscopic assessment of the shoulder, patients that have a confirmed irreparable tear will be randomized into one of two groups: arthroscopic partial repair or superior capsular reconstruction. Surgical techniques will be standardized. Allocation will be concealed using a centralized 24-hour computerized randomization system that will allow Internet-based allocation. A random number generator will be used to create a 1:1 allocation scheme for randomization of the patient into one of the two treatment groups. The post-operative therapy regimen will be the same for each group.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic shoulder pain and/ or weakness (regardless of baseline range of motion/ psuedoparalysis)
* Massive rotator cuff tear, identified by MRI as being greater than 4 cm in greatest diameter, and involvement of the entire supraspinatus and infraspinatus.
* Failure of at least a 3 month trial of non-surgical treatment including physiotherapy and activity modifications
* Irreparable tear determined intra-operatively using standard arthroscopic techniques
* Informed consent obtained

Exclusion Criteria:

* Absence of subscapularis muscle insertion, or irreparable subscapularis tear
* Advanced rotator cuff tear arthropathy (Hamada Grade 3+) or glenohumeral osteoarthritis (Samilson-Prieto grade 2+)
* Acute tears (within 6 months)
* Neurologic injury causing paralysis of affected shoulder / arm
* Any previous surgery to the affected shoulder
* Limited life expectancy due to significant medical co-morbidity or medical contraindication to surgery (ASA Grade IV or higher)
* Anticipated problems with ability to maintain follow-up in the judgement of the investigators (ie. patients with no fixed address, etc.)
* Are there any non-orthopedic comorbidities that put the patient at significant risk?

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The American Shoulder and Elbow Surgeons Shoulder Score (ASES) | 1 year post operative
  Functional Outcome Score
  Sub scales: Pain (10 cm VAS); function/disability (10 items, each rated on 4-point Likert scale for level of difficulty)
  Score range: Pain subscale 0-50 ASES points; function/disability subscale 0-50 ASES points. Total score 0-100 ASES points (0 = worse pain and functional loss/disability)

SECONDARY OUTCOMES:
Complication rate | 1 year post operative
  Incidence of minor and major complications related to each procedure.
Recruitment rate | 1 year post operative
  Assessment of number of eligible patients identified and number enrolled and randomized.
Constant-Murley Score | 1 year post operative
  Functional outcome score
  Sub scales: Pain item (4 Likert levels), Activities of Daily Living (Likert scales), Mobility (2 points for every 30 degrees of elevation), Strength (1 point per 0.5 kg)
  Score Range: pain (0-15 points), activities of daily living (0-20 points), strength (0-25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (0-40 points). Total score: 0-100. The higher the score, the higher the quality of the function.
Western Ontario Rotator Cuff Index | 1 year post operative
  Functional outcome score
  Consists of 21 visual analog scale (VAS) items organised in 5 subscales: physical symptoms, sports/recreation, work, lifestyle, and emotions.
  Each item in WORC has a possible score from 0-100 (100mm VAS). Scores can be computed for individual subscales and summated for a total score, which can range from 0-2100, with a higher score representing lower quality of life.
Pain: Numeric Rating Scale | 1 year post operative
  Scale range: 0 to 10 (whole number integers). Higher scores represent more pain.
Range of Motion | 1 year post operative
  Measured by handheld goniometer
EQ-5D | 1 year post operative
  Health Related Quality of Life
  The EQ-5D questionnaire is made up for two components; health state description and evaluation.
  In description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3.
  Visual analogue scale: 20 cm vertical scale with end points of 0 and 100. 0 corresponds to " the worst health you can imagine", and 100 corresponds to "the best health you can imagine".
Xray: Acromio-Humeral Interval | 1 year post operative
  Measured distance from inferior acromion to superior humeral head at the closest distance. Distance in millimetres.
Xray: Degenerative Change | 1 year post operative
  Measured by Samilson-Prieto Grade:
  Mild Arthritis (Grade 1): inferior humeral and/or glenoid exostosis < 3mm in height
  Moderate Arthritis (Grade 2): inferior humeral and/or glenoid exostosis measuring 3mm to 7mm slight gleno-humeral irregularity
  Severe Arthritis (Grade 3): inferior humeral and/or glenoid exostosis measuring > 7mm gleno-humeral joint narrowing and sclerosis
MRI - graft healing | 1 year post operative
  Assess graft integrity: Healed or Torn
MRI - tear size | 1 year post operative
  Assess size of recurrent tear (in maximum anterior to posterior and medial to lateral dimensions). Measured in cm.
MRI - fatty degeneration | 1 year post operative
  Measured by Goutallier classification of each rotator cuff muscle:
  grade 0: normal muscle grade 1: some fatty streaks grade 2: less than 50% fatty muscle atrophy grade 3: 50% fatty muscle atrophy grade 4: greater than 50% fatty muscle atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Henry, MD, FRCSC, Principal Investigator — Sunnybrook Health Sciences
Locations (2):
- Canada (2):
  - Sunnybrook Holland Orthopaedic & Arthritic Centre, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No